CLINICAL TRIAL: NCT06243536
Title: The Effect of Semaglutide on Disordered Eating Behaviour in Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Collaborators: University of Zagreb School of Medicine (Unknown)
Responsible Party: Principal Investigator, Jelena Marinkovic Radosevic, Principal Ivenstigator, University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 251-29-1 1/3-23-06
Record Dates: First submitted 2024-01-13; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes; Overweight; Disordered Eating Behaviors
Keywords: Randomized controlled trial; Semaglutide; Incretin hormones; Glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Disordered Eating Behavior | interventions — semaglutide; Standard of Care; Metformin; Sulfonylurea Compounds; Pioglitazone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Type 2 diabetic patients without disordered eating behaviour (Placebo Comparator): Treated with standard of care.
  Interventions: Drug: standard of care
- Type 2 diabetic patients with disordered eating behaviour A (Placebo Comparator): Treated with standard of care.
  Interventions: Drug: standard of care
- Type 2 diabetic patients with disordered eating behaviour B (Experimental): Receiving semaglutide for 12 weeks
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Semaglutide will be administered through 12 weeks.
  Arms: Type 2 diabetic patients with disordered eating behaviour B
Drug: standard of care — Patients not assigned to receive semaglutide will receive standard of care.
  Other Names: Metformin, Sulfonylureas, Sodium-glucose cotransporter-2 inhibitors, pioglitazone
  Arms: Type 2 diabetic patients with disordered eating behaviour A; Type 2 diabetic patients without disordered eating behaviour

SUMMARY:
The aim of this study is to evaluate the effect of glucagon-like peptide-1 (GLP-1) receptor agonist semaglutide on disordered eating behaviour in patients with overweight and type 2 diabetes. The investigators will also evaluate serum concentrations of incretin hormones GLP-1 and glucose-dependent insulinotropic polypeptide (GIP), as well as glucose variability using continuous glucose monitoring (CGM) devices before and after semaglutide, and determine his influence on eating disorders.

In this prospective study the investigators aim to recruit 60 patients with type 2 diabetes and randomize them based on the presence of a disordered eating behaviour diagnosed by a validated questionnaire (1:1). Patients with a disordered eating behaviour will further be randomized (1:1) to receive semaglutide. At baseline and after 12 weeks of semaglutide therapy, the investigators will reevaluate glucose variability over 14 days using a continuous glucose monitoring device (CGM).

With this study the investigators will determine the impact of GLP-1 receptor agonist semaglutide on disordered eating behaviour in patients with overweight and type 2 diabetes. This study will contribute to the knowledge about the role of incretin hormones and glucose variability in eating disorders in this population of patients.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted in Clinical Hospital Center Sestre milosrdnice and University of Zagreb School of medicine. Patients will be randomized after completing the EAT-26 questionnaire (1:1), in group with disordered eating behaviour (n=30) if participants scored >20 points, and group without disordered eating behaviour (n=30) if participants scored ≤20 points. Group of patients with disordered eating behaviour will be further randomized whether participants will receive semaglutide (n=15) with standard care or if participants will be treated with standard care (n=15). The investigators will evaluate baseline EAT-26 score, GLP-1 and GIP blood levels in a mixed meal test, anthropometric measurements (weight, BMI, waist circumference), biochemical parameters (complete blood count, glucose, insulin, c-peptide, HbA1c, urea, creatinine, uric acid, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), international normalized ratio (INR), albumin, serum lipid levels (cholesterol. HDL, LDL, triglyceride), C reactive protein (CRP), urine sediment and their changes at the end of the trial (except mixed meal test). Also, through 14 days at the beginning and 14 days before the end of the trial, patients will keep a food diary and have intermittently scanned continuous glucose monitor (FreeStyle Libre Pro CGM device, Abbott).

A factor analysis of EAT-26 scores will be conducted to form 3 (expected) latent variables (components). To assess the effect on dietary habits, the difference in EAT-26 total score and latent variables between subjects randomized to semaglutide and control subjects (randomized to standard care) will be assessed after 3 months of treatment. The data will be analysed in a general linear model, with basal covariates: age, sex, BMI and score at the beginning of treatment. In the same way, the effect of semaglutide on GLP1 concentrations (basal covariate: basal concentration next to the location of the EAT-26 score) will be evaluated, separately for the condition before and after the mixed meal test. GLP-1 and GIP concentrations will be compared between subjects with ("exposed") and without (control) eating disorders, in a generalized linear model for repeated measurements (GLP-1 concentration before and after mixed meal test) with fixed covariates: age, sex, BMI, time ( before or after mixed meal test) and exposure*time interactions. Type I (α) error=0.05.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes, age 18-65, BMI ≥28 kg/m2, HbA1c>7%, glp-1 receptor agonist naïve

Exclusion Criteria:

* hepatic impairment (Child Pugh score C), renal impairment (eGFR<30 ml/min), use of medication that affect eating (GLP-1 receptor agonists, antidepressants, antiobesity medications, glucocorticoids, insulin, oral contraceptives, hormonal therapy), conditions that can affect eating (hypothyroidism, hyperthyroidism, Cushing syndrome, acromegaly, adrenal insufficiency, pregnancy, breastfeeding), contraindications for semaglutide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Eating Attitude Test (EAT-26) questionnaire score | EAT-26 questionnaire will be assessed at the beginning of the trial and at the end of the trial after 12 weeks.
  Investigate the effect of semaglutide on the intensity of disordered eating behaviour quantified by the EAT-26 questionnaire in patients with overweight and type 2 diabetes. Possible scores in EAT-26 questionnaire min.0-max 78, with lower score indicating better outcome.

SECONDARY OUTCOMES:
Continuous glucose monitoring parameter (Glycemic Variability) | CGM parameter will be assessed through 14 days at the beginning of the trial and through 14 days at the end of the trial after 12 weeks.
  Investigate the effect of semaglutide on continuous glucose monitoring parameter glycemic variability defined by the measurement of fluctuations of glucose over a given interval of time (14 days) presented as coefficient of variation (CV) with values of %CV ≥ 36, as high glycemic variability.
Concentration of incretin hormones (GLP-1, GIP) | At the beginning of the trial (before semaglutide administration)
  To assess the concentrations of incretin hormones (GLP-1, GIP) in group of participants with eating behaviour disorder and in group of participants without eating behaviour disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Osmanović Barilar, Professor, Study Chair — University of Zagreb School of Medicine
Locations (1):
- UH Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Nieto-Martinez R, Gonzalez-Rivas JP, Medina-Inojosa JR, Florez H. Are Eating Disorders Risk Factors for Type 2 Diabetes? A Systematic Review and Meta-analysis. Curr Diab Rep. 2017 Nov 22;17(12):138. doi: 10.1007/s11892-017-0949-1. PMID 29168047
- [Background] Garcia-Mayor RV, Garcia-Soidan FJ. Eating disoders in type 2 diabetic people: Brief review. Diabetes Metab Syndr. 2017 Jul-Sep;11(3):221-224. doi: 10.1016/j.dsx.2016.08.004. Epub 2016 Aug 22. PMID 27575047
- [Background] Presseller EK, Patarinski AGG, Zhang F, Page KA, Srivastava P, Manasse SM, Juarascio AS. Glucose variability: A physiological correlate of eating disorder behaviors among individuals with binge-spectrum eating disorders. Int J Eat Disord. 2022 Dec;55(12):1788-1798. doi: 10.1002/eat.23838. Epub 2022 Oct 28. PMID 36305323
- [Background] Suh S, Kim JH. Glycemic Variability: How Do We Measure It and Why Is It Important? Diabetes Metab J. 2015 Aug;39(4):273-82. doi: 10.4093/dmj.2015.39.4.273. PMID 26301188
- [Background] Papelbaum M, de Oliveira Moreira R, Coutinho WF, Kupfer R, Freitas S, Raggio Luz R, Appolinario JC. Does binge-eating matter for glycemic control in type 2 diabetes patients? J Eat Disord. 2019 Sep 6;7:30. doi: 10.1186/s40337-019-0260-4. eCollection 2019. PMID 31516703
- [Background] Martinez M, Santamarina J, Pavesi A, Musso C, Umpierrez GE. Glycemic variability and cardiovascular disease in patients with type 2 diabetes. BMJ Open Diabetes Res Care. 2021 Mar;9(1):e002032. doi: 10.1136/bmjdrc-2020-002032. PMID 33762313
- [Background] Daly A, Hovorka R. Technology in the management of type 2 diabetes: Present status and future prospects. Diabetes Obes Metab. 2021 Aug;23(8):1722-1732. doi: 10.1111/dom.14418. Epub 2021 May 20. PMID 33950566
- [Background] Mancuso SG, Newton JR, Bosanac P, Rossell SL, Nesci JB, Castle DJ. Classification of eating disorders: comparison of relative prevalence rates using DSM-IV and DSM-5 criteria. Br J Psychiatry. 2015 Jun;206(6):519-20. doi: 10.1192/bjp.bp.113.143461. Epub 2015 Mar 5. PMID 25745131
- [Background] Nicolau J, Simo R, Sanchis P, Ayala L, Fortuny R, Zubillaga I, Masmiquel L. Eating disorders are frequent among type 2 diabetic patients and are associated with worse metabolic and psychological outcomes: results from a cross-sectional study in primary and secondary care settings. Acta Diabetol. 2015 Dec;52(6):1037-44. doi: 10.1007/s00592-015-0742-z. Epub 2015 Apr 5. PMID 25841588
- [Background] Herpertz S, Albus C, Kielmann R, Hagemann-Patt H, Lichtblau K, Kohle K, Mann K, Senf W. Comorbidity of diabetes mellitus and eating disorders: a follow-up study. J Psychosom Res. 2001 Nov;51(5):673-8. doi: 10.1016/s0022-3999(01)00246-x. PMID 11728508
- [Background] Watts AG, Kanoski SE, Sanchez-Watts G, Langhans W. The physiological control of eating: signals, neurons, and networks. Physiol Rev. 2022 Apr 1;102(2):689-813. doi: 10.1152/physrev.00028.2020. Epub 2021 Sep 6. PMID 34486393
- [Background] Tong J, D'Alessio D. Eating disorders and gastrointestinal peptides. Curr Opin Endocrinol Diabetes Obes. 2011 Feb;18(1):42-9. doi: 10.1097/MED.0b013e328341e12b. PMID 21157325
- [Background] Smith KR, Moran TH. Gastrointestinal peptides in eating-related disorders. Physiol Behav. 2021 Sep 1;238:113456. doi: 10.1016/j.physbeh.2021.113456. Epub 2021 May 11. PMID 33989649
- [Background] Dixon KN, O'Dorisio TM, Zipf W, Cataland S. Gastric inhibitory polypeptide (GIP) in anorexia nervosa. Int. J. Eat. Disord. 1985, 4: 597-604
- [Background] Cho YM, Fujita Y, Kieffer TJ. Glucagon-like peptide-1: glucose homeostasis and beyond. Annu Rev Physiol. 2014;76:535-59. doi: 10.1146/annurev-physiol-021113-170315. Epub 2013 Nov 13. PMID 24245943
- [Background] Elliott RM, Morgan LM, Tredger JA, Deacon S, Wright J, Marks V. Glucagon-like peptide-1 (7-36)amide and glucose-dependent insulinotropic polypeptide secretion in response to nutrient ingestion in man: acute post-prandial and 24-h secretion patterns. J Endocrinol. 1993 Jul;138(1):159-66. doi: 10.1677/joe.0.1380159. PMID 7852887
- [Background] Sharma D, Verma S, Vaidya S, Kalia K, Tiwari V. Recent updates on GLP-1 agonists: Current advancements & challenges. Biomed Pharmacother. 2018 Dec;108:952-962. doi: 10.1016/j.biopha.2018.08.088. Epub 2018 Sep 27. PMID 30372907
- [Background] Nauck MA, Quast DR, Wefers J, Meier JJ. GLP-1 receptor agonists in the treatment of type 2 diabetes - state-of-the-art. Mol Metab. 2021 Apr;46:101102. doi: 10.1016/j.molmet.2020.101102. Epub 2020 Oct 14. PMID 33068776
- [Background] Baggio LL, Drucker DJ. Biology of incretins: GLP-1 and GIP. Gastroenterology. 2007 May;132(6):2131-57. doi: 10.1053/j.gastro.2007.03.054. PMID 17498508
- [Background] Tommerdahl KL, Nadeau KJ, Bjornstad P. Mechanisms of Cardiorenal Protection of Glucagon-Like Peptide-1 Receptor Agonists. Adv Chronic Kidney Dis. 2021 Jul;28(4):337-346. doi: 10.1053/j.ackd.2021.06.001. PMID 34922690
- [Background] Bullock BP, Heller RS, Habener JF. Tissue distribution of messenger ribonucleic acid encoding the rat glucagon-like peptide-1 receptor. Endocrinology. 1996 Jul;137(7):2968-78. doi: 10.1210/endo.137.7.8770921.
- [Background] Drucker DJ. Mechanisms of Action and Therapeutic Application of Glucagon-like Peptide-1. Cell Metab. 2018 Apr 3;27(4):740-756. doi: 10.1016/j.cmet.2018.03.001. PMID 29617641
- [Background] Hsu TM, Noble EE, Liu CM, Cortella AM, Konanur VR, Suarez AN, Reiner DJ, Hahn JD, Hayes MR, Kanoski SE. A hippocampus to prefrontal cortex neural pathway inhibits food motivation through glucagon-like peptide-1 signaling. Mol Psychiatry. 2018 Jul;23(7):1555-1565. doi: 10.1038/mp.2017.91. Epub 2017 May 2. PMID 28461695
- [Background] McElroy SL, Mori N, Guerdjikova AI, Keck PE Jr. Would glucagon-like peptide-1 receptor agonists have efficacy in binge eating disorder and bulimia nervosa? A review of the current literature. Med Hypotheses. 2018 Feb;111:90-93. doi: 10.1016/j.mehy.2017.12.029. Epub 2018 Jan 2. PMID 29407005
- [Background] Robert SA, Rohana AG, Shah SA, Chinna K, Wan Mohamud WN, Kamaruddin NA. Improvement in binge eating in non-diabetic obese individuals after 3 months of treatment with liraglutide - A pilot study. Obes Res Clin Pract. 2015 May-Jun;9(3):301-4. doi: 10.1016/j.orcp.2015.03.005. Epub 2015 Apr 11. PMID 25870084
- [Background] Jensterle M, Kocjan T, Kravos NA, Pfeifer M, Janez A. Short-term intervention with liraglutide improved eating behavior in obese women with polycystic ovary syndrome. Endocr Res. 2015;40(3):133-8. doi: 10.3109/07435800.2014.966385. Epub 2014 Oct 20. PMID 25330463
- [Background] Da Porto A, Casarsa V, Colussi G, Catena C, Cavarape A, Sechi L. Dulaglutide reduces binge episodes in type 2 diabetic patients with binge eating disorder: A pilot study. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):289-292. doi: 10.1016/j.dsx.2020.03.009. Epub 2020 Mar 31. PMID 32289741
- [Background] Frias JP, Nakhle S, Ruggles JA, Zhuplatov S, Klein E, Zhou R, Strange P. Exenatide once weekly improved 24-hour glucose control and reduced glycaemic variability in metformin-treated participants with type 2 diabetes: a randomized, placebo-controlled trial. Diabetes Obes Metab. 2017 Jan;19(1):40-48. doi: 10.1111/dom.12763. Epub 2016 Sep 21. PMID 27527911
- [Background] FLAT-SUGAR Trial Investigators. Glucose Variability in a 26-Week Randomized Comparison of Mealtime Treatment With Rapid-Acting Insulin Versus GLP-1 Agonist in Participants With Type 2 Diabetes at High Cardiovascular Risk. Diabetes Care. 2016 Jun;39(6):973-81. doi: 10.2337/dc15-2782. Epub 2016 Apr 19. PMID 27208320
- [Background] Pratley RE, Catarig AM, Lingvay I, Viljoen A, Paine A, Lawson J, Chubb B, Gorst-Rasmussen A, Miresashvili N. An indirect treatment comparison of the efficacy of semaglutide 1.0 mg versus dulaglutide 3.0 and 4.5 mg. Diabetes Obes Metab. 2021 Nov;23(11):2513-2520. doi: 10.1111/dom.14497. Epub 2021 Aug 9. PMID 34286894
- [Background] Takahashi Y, Nomoto H, Yokoyama H, Takano Y, Nagai S, Tsuzuki A, Cho KY, Miya A, Kameda H, Takeuchi J, Taneda S, Kurihara Y, Atsumi T, Nakamura A, Miyoshi H; SWITCH-SEMA 1 study group. Improvement of glycaemic control and treatment satisfaction by switching from liraglutide or dulaglutide to subcutaneous semaglutide in patients with type 2 diabetes: A multicentre, prospective, randomized, open-label, parallel-group comparison study (SWITCH-SEMA 1 study). Diabetes Obes Metab. 2023 Jun;25(6):1503-1511. doi: 10.1111/dom.14998. Epub 2023 Feb 28. PMID 36722623
- [Background] Rahelic D, Altabas V, Bakula M, Balic S, Balint I, Markovic BB, Bicanic N, Bjelinski I, Bozikov V, Varzic SC, Car N, Berkovic MC, Orlic ZC, Deskin M, Sunic ED, Tomic NG, Goldoni V, Gradiser M, Mahecic DH, Balen MJ, Erzen DJ, Majanovic SK, Kokic' S, Krnic M, Kruljac I, Liberati-Cizmek AM, Martina L, Metelko Z, Mirosevic G, Vrbica SM, Renar IP, Petric D, Prasek M, Prpic-Kizevac I, Radman M, Soldo D, Saric T, Tesanovic S, Kurir TT, Wensveen TT, Botica M, Vrkljan M, Rotkvic VZ, Zoric C, Krznaric Z. [CROATIAN GUIDELINES FOR THE PHARMACOTHERAPY OF TYPE 2 DIABETES]. Lijec Vjesn. 2016 Jan-Feb;138(1-2):1-21. Croatian. PMID 27443001
- [Background] Meier JJ. Efficacy of Semaglutide in a Subcutaneous and an Oral Formulation. Front Endocrinol (Lausanne). 2021 Jun 25;12:645617. doi: 10.3389/fendo.2021.645617. eCollection 2021. PMID 34248838
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] Ambrosi-Randic N, Pokrajac-Bulian A. Psychometric properties of the eating attitudes test and children's eating attitudes test in Croatia. Eat Weight Disord. 2005 Dec;10(4):e76-82. doi: 10.1007/BF03327495. PMID 16682865
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- See also: Magliano DJ, Boyko EJ; IDF Diabetes Atlas 10th edition scientific committee. IDF diabetes atlas 10th ed. [Internet]. Brussels: International Diabetes Federation; 2021 — http://diabetesatlas.org
- See also: Buble T, Čavlina M. Nacionalni registar osoba sa šećernom bolešću CroDiab. Izvješće za 2022. [Internet]. Zagreb: Hrvatski zavod za javno zdravstvo; 2022 — https://www.hzjz.hr/wp-content/uploads/2023/03/Izvjesce_za_2022_godinu.pdf
- See also: U. S. Department of Agriculture, Agricultural Research Service. USDA National Nutrient Database for Standard Reference, Legacy Release. [Internet]. 2018 — http://www.ars.usda.gov/nutrientdata